CLINICAL TRIAL: NCT07091565
Title: SPARC: Supporting Sexual Recovery in Women With Bladder Cancer
Brief Title: Supporting Sexual Recovery in Women With Bladder Cancer
Acronym: SPARC
Status: Enrolling by invitation | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's & St Thomas' NHS FT (Unknown); The Royal Marsden NHS FT (Unknown); Sheffield Teaching Hospitals NHS FT (Unknown)
Responsible Party: Sponsor
Other Study IDs: 335939
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Cystectomy; Female Sexual Dysfunction
Keywords: Bladder cancer; transitional cell carcinoma; radical cystectomy; anterior exenteration; exenteration; sexual function; women; female; gynaecological organs
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Experienced patients
  Interventions: Other: Qualitative interview/Focus group
- HCP: Experienced healthcare professionals
  Interventions: Other: Qualitative interview/Focus group

INTERVENTIONS:
Other: Qualitative interview/Focus group — Participants will take part in a 1:1 interview or focus group

SUMMARY:
This study looks at how bladder cancer and removing the bladder can affect women's sexual well-being. Bladder cancer can be more serious in women, and treatment like bladder removal can impact how they feel about themselves and their relationships. Women who've gone through this say it's important to talk about and get support for their sexual recovery.

The study has three main parts. First, it reviews what is already known. Next, it involves talking to women with bladder cancer and the doctors and nurses who care for them. Finally, the team will use what they learn to create a toolkit to help healthcare workers support women's sexual recovery.

Women with bladder cancer are helping to design this study. Their input shapes the questions and tools. The final toolkit will include training for doctors and nurses and be shared online and through charities. The aim is to make this part of regular healthcare.

DETAILED DESCRIPTION:
Background & Aims Bladder cancer is one of the top ten cancers in the UK. In women, it can be more aggressive, meaning it can be more harmful. Bladder cancer often needs invasive treatment or procedures such as bladder removal. This can cause problems with a woman's sexual well-being and recovery.

There are different types of bladder cancer, and each requires a different treatment. In high-risk types, a more intensive treatment is required. The patient may need to have their bladder removed. The bladder is replaced with an alternative option for urine drainage such as a bag on the skin. In bladder removal, evidence tells us that there will be an impact on a woman's sexual well-being.

Sexual recovery is an important aspect of personal wellbeing and quality of life after cancer treatment. We have worked with women to develop this proposal and they tell us this is important to them.

This study aims to examine this aspect of well-being in women with bladder cancer and having bladder removal. The study will develop a toolkit alongside women to support sexual recovery in this group of patients.

What will the study involve? The study has been designed in stages to breakdown the individual elements.

Stage 1:

The initial stage involves a detailed examination of the existing literature to understand what needs to be discovered.

Stage 2:

The next stage requires in-depth investigation through interviewing patients individually or in a group. Doctors and nurses will also be interviewed about sexual well-being and bladder cancer. Findings from these interviews will be looked at to identify common themes and to understand how care is given.

Stage 3:

Findings from Stages 1 and 2 will be used to co-design a toolkit. The toolkit will be designed in partnership with patients and clinical experts.

It is anticipated that the toolkit will involve education sessions face to face or online to allow the healthcare provider to give better care. The toolkit will be tested to check it is meeting the needs of patients and that it is acceptable to users.

Public Involvement and Engagement This is a co-design project. This means that patients are involved in the project at every stage. At the start, a project codesign group has been created. This includes five patients with experience of bladder cancer. The group is from different backgrounds and further efforts will be made to include people from under-represented groups. For example, the patient group thought it was important for patients to be offered interviews alone or in groups. This was particularly important for the members from under-represented groups, so the study design was amended.

Considerations Prior to starting, ethical approval will be sought to be sure the study will not cause harm. Patients will be invited to participate by post or email. Participation will be voluntary and can be withdrawn. Recruited patients will be allocated an anonymous identification code and all data will be stored in a safe way. Some participants may feel upset during the study and need extra support. If this happens, they will be referred for specialist help.

Outcomes A toolkit will be designed for healthcare professionals. The toolkit will help healthcare professionals to support women's sexual recovery. The toolkit will be tested to make sure it works. The findings will be shared with patients online and through charity groups. This will be achieved through explanatory animations. Doctors and nurses will be encouraged to complete the training and will be alerted to it at professional meetings and groups. The final aim is to include this toolkit within clinical training and guidelines.

ELIGIBILITY:
Patient Inclusion

* All women and other patients with a clitoris, vagina, neo-vagina or neo-clitoris
* Have a diagnosis of BCa-any grade/stage and have had a cystectomy (bladder removal)
* At least 6 months after cystectomy
* >/ 18 years old
* Written informed consent.

HCP Inclusion

* All those working directly within a bladder cancer speciality
* Professional registration
* Written informed consent

Patient Exclusion

* Poor command of the English language to the extent that the researcher judges this to critically undermine the ability to achieve the objectives of the interview.
* A judgement by the researcher or the individual's clinician, based on either clinical appraisal (capacity assessment) or review of the individual's medical notes, that the individual has a cognitive functioning impairment that would interfere with ability to understand and complete the interview.
* Documentation in the accessible medical notes of a psychiatric condition that would hamper participation in interview.
* A judgement by the researcher or the individual's clinician, based on either clinical appraisal or review of the individual's medical notes, that the individual is too ill to participate; or is ill enough that participation would produce an unreasonable burden on that individual.
* Aged <18 years.

HCP Exclusion:

-Those without professional registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female bladder cancer patients who have undergone bladder removal.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Qualitative only | 01/08/25-01/06/26
  Thematic analysis following an inductive framework approach to elicit codes and themes from the interviews.

SECONDARY OUTCOMES:
Intervention development | 06/2026-06/2027
  Emerging codes and themes from the qualitative interviews will inform intervention design and intervention development.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No